CLINICAL TRIAL: NCT03677284
Title: Managing Time With Dementia: Effects of Time Assistive Products on Time-processing Ability, Daily Time Management and Well-being in People With Dementia
Brief Title: Managing Time With Dementia: Effects of Time Assistive Products in People With Dementia
Acronym: MTD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Dalarna University (Other); Manipal University (Other); National Rehabilitation Center for Persons with Disabilities, Japan (Other)
Responsible Party: Principal Investigator, Gunnel Janeslätt, PhD, Principal Investigator, Occupational Therapist (reg), Researcher, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: FORTE 2017-00029
Record Dates: First submitted 2018-08-20; First posted 2018-09-19 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Dementia
Keywords: Intervention study; Assistive products; Elderly people
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Assessments at baseline (t1) is done for each person with dementia (PwD) with informed consent. The coding of each PwD is determined by the memory clinic (first two digits in the code, 10 - 70) and consecutive starting with 01 and on.
  A stratified randomization will be prepared in advance by the researchers, in closed envelopes, for each memory clinic. When the assessment is done, the occupational therapist opens the top envelope marked with the code of the PwD to find out allocation to intervention or control.
  Intervention will be provided by the occupational therapist at the memory clinic or at other out-patient service during three months. The second data collection (t2) will be done by research assistants. After the assessment (t2), the control group will be offered intervention with prescribed time assistive products, followed by a third assessment (t3) after another three months (6 months after baseline).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The assessments at three and six months (for intervention group t2, for control group t2 and t3) will be performed by research assistants to avoid bias from the care providers (occupational therapists giving intervention). It is anticipated that the research assistant will not be informed of what group the PwD was allocated to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Information brochure about daily time management, frequent problems, and suggested strategies to manage them.
  Time assistive product. Time assistive products for time perception are products making the passage of time visible and understandable, to know for how long to perform an activity or how long to wait until the next activity starts e.g a time log.
  Time assistive products for time orientation includes the use of schedules, calendars and other visual aids to promote orientation to the time of the day, week, or year.
  Time assistive products for time management would compensate for deficits in time management and focus on self-scheduling skills.
  Interventions: Other: Time assistive products; Other: Information brochure
- Control group (Active Comparator): Information brochure about daily time management, frequent problems, and suggested strategies to manage them.
  Interventions: Other: Information brochure

INTERVENTIONS:
Other: Time assistive products — The decision on the specific time assistive product to be prescribed will be decided based on current knowledge and the personal goal of the PwD.
  Arms: Intervention group
Other: Information brochure — The information brochure will provide information frequent problems about daily time management and suggest strategies to manage them.

SUMMARY:
Sweden, like most countries, is undergoing population ageing. This is accompanied by an epidemiologic transition of equal importance, leading to a greater number of people than ever before affected by dementia. Dementia affects thinking, memory, behavior and ability to perform everyday activities, including daily time management. Time orientation and daily management has been shown to influence well-being in older people. There is evidence suggesting that time assistive products can have positive effects on the well-being of both primary users and informal care givers, but this is not sufficient to provide evidence-based guidance for effective interventions, nor to develop innovative and effective solutions.

In order to contribute to the development and use of affordable and appropriate innovative assistive products and services for older people with mild or moderate dementia, the purposes of this project are to investigate and model the relationship between the use of time assistive products by older people with dementia, their daily time management and their well-being, and to devise strategies for the acceptance and use of such products by older people with dementia and informal caregivers.

A mixed longitudinal approach will be used to attain the first purpose, while the second purpose will be accomplished by applying a qualitative method. Women and men aged 65 or older diagnosed with early or moderate dementia (n=74), and their significant others will be eligible for inclusion.

Cooperation with researchers in India and Japan will generate a set of core data, which allows for cross-cultural comparisons of factors related to daily time management and well-being. The three-year project started September 2017, the main study in September 2018.

This project can be expected to contribute important knowledge that can advance the effectiveness of cornerstone social policies such as support for ageing in place and healthy and active ageing, and the reduction of social exclusion of older people.

DETAILED DESCRIPTION:
Introduction

How time is managed is of great importance for daily life, including participation and well-being (Christiansen, 2005). Time management behaviors relate positively to perceived control of time, satisfaction and health, and negatively to stress (Claessens, van Eerde, Rutte, & Roe, 2007). Prenda and Lachman (2001) demonstrated that planning predicted life satisfaction in older people, while Ouwehand et al. (2006) found that future time orientation was important for their well-being. The capacity for concrete planning has also been shown to predict well-being in older people over a one-year period (Tovel & Carmel, 2014). More broadly, the capacity to orient in time and plan is essential in goal-setting, the benefits of which have been extensively documented in older people (Frazier, Newman, & Jaccard, 2007).

Sweden, like most countries, is undergoing population ageing and an epidemiologic transition, which is leading to a greater number of people than ever before affected by dementia. Caused by a variety of brain illnesses, dementia affects thinking, memory, behavior and ability to perform everyday activities, including daily time management. Time perception and time orientation are essential functions that are compromised in dementia (El Haj, Gandolphe, Wawrziczny, & Antoine, 2016; Grewal, 1995; Iwamoto & Hoshiyama, 2012).Temporal relationships, and the coherence of past, present and future become unclear and vague; past time disappears and planning for the future seems less important or impossible. People with dementia may experience difficulties with regard to knowing, remembering and planning "when", and knowing "how long" different activities or situations would last. This causes problems to plan and keep appointments. Moreover, not being able to judge the length of time intervals can make them feel lonely when their spouse or informal caregiver is away due to a failure to gauge the length of the absence, which can cause stress and worry for both the person with dementia (PwD) and the caregiver (Nygard & Johansson, 2001)

Appropriate and effective assistive products can offer PwD and their relatives the opportunity to develop a more mutually satisfactory care relationship and enhance the person with dementia's capacity for self-management. Then, the time spent with the family caregiver is not reduced to a succession of required care tasks but can encompass more meaningful social and emotional engagements.

A review of technology for older people with cognitive or other impairments concluded that the cost-benefit was generally high or very high (Dahlberg, 2014). Despite this, the uptake of assistive products is quite low because of lack of competence, awareness, organization, user training and reliability of technical solutions. Family caregivers played a significant role in whether or not assistive products were absorbed into the everyday life practice (Arntzen, Holthe, & Jentoft, 2014). Moreover, it is important that assistive products are easy to maintain and fit into the context of use in order to increase the sense of control of the products by users with dementia, and thereby promote the goal achievement and usability of the products (Lindqvist, Larsson, & Borell, 2015). Research has also highlighted the necessity of adaptation of the products to individual users, regardless whether they are mainstream or specially-designed products (Boman, Nygård, & Rosenberg, 2014; Boman, Persson, & Bartfai, 2016).

To facilitate daily time management of people with cognitive impairments, time assistive products have been developed and evaluated (Gillespie, Best, & O'Neill, 2012). Enhanced time management in a PwD, with improved time keeping, planning capacity and goal-setting, could increase the potential for social interaction and participation, while reducing the negative impact and increasing the positive value of caregiving for relatives as identified in Balducci et al. (2008). It has been reported that assistive products can support people with dementia to orientate to dates, weekdays and time; to go back to sleep at night; to feel calmer, in control and more secure; and to cope and manage more effectively and to carry out daily routines. The products can increase the ability of people with dementia to retain roles, reduce the need for them to ask others about day and time, and reduce the number of times they wake up others at night. This helps caregivers to have better sleep and feel relieved, and to have a less stressful relation with the primary user of the product (Forsenäs et al. 2011; Hagen 2006)(Holthe, Hagen, Bjørneby, & Vollgate, 1998; Topo et al., 2007). Assistive products can provide users with an overview of the day, and remind them about activities (e.g., meals, medicine, visits and training). They can also give them time to do other things between scheduled activities, and inform about time and date (Bakken 2014). It has also been reported that assistive products can save time and effort, decrease worries and stress, and increase a sense of safety, which enabled users with dementia to perform their valued activities (Lindqvist, Nygård, & Borell, 2013). Still, although daily time management is such a significant difficulty in dementia, the evidence from populations with dementia is limited in both quantity and quality.

It is of vital importance to implement a research project that creates knowledge for developing effective time-related interventions for improving the well-being of people with dementia and informal caregivers.

Purposes

In order to contribute to the development and use of affordable and appropriate innovative assistive technology for daily time management among older people with dementia, the purposes of this project are:

* to investigate and model the relationship between the use of time assistive products by older people with mild to moderate dementia, their daily time management and their well-being, and
* to devise strategies for the acceptance and use of such products by older people with dementia and informal caregivers.

The purposes of this project are relevant in the field of ageing and health. The first purpose will explore how supportive technologies for functional abilities (in the form of time assistive products) affect older people's daily time management and well-being (including, activities, participation and independence). In addition to providing evidence of the effects of the products, the first purpose will result in an empirically based theoretical model to better understand their role. This model will offer a basis for the development of new and improved products and services.

The second purpose will contribute knowledge of experiences in PwD directly and via their informal caregiver, about their use of time assistive products and their perceptions of learning how to use them. This includes identifying features that need to be integrated in the design of products and services in order to effectively address the needs of older PwD and their informal caregivers. This purpose will also contribute to the development of new and improved products and services by devising strategies that consider current barriers to and facilitators of the acceptance and use of such products.

The project will investigate time assistive devices for people with dementia from three perspectives - occupational therapists, PwDs and their informal caregivers. This is done in three phases with the following research questions:

Research questions

Phase I - The perspective of occupational therapists:

1. What are the occupational therapist's experiences of prescribing time assistive products for persons with mild or moderate dementia, focusing on facilitating and hindering factors?

Phase II - Intervention with focus on persons with mild or moderate dementia and their informal caregivers:

2a) To what degree can time assistive products support persons with mild or moderate dementia in reaching their personal activity goals, in performance of daily activities and in satisfaction with the performance? 2b) What is the relation between time-processing ability, daily time management, and well-being of people with mild or moderate dementia within differing socioeconomic and care contexts? 2c) How can intervention with time assistive products affect time-processing ability, daily time management and well-being of people with dementia and the well-being of their informal caregivers? 2d) Are there differences in results of research questions 2a - 2c between different cultures (Sweden, India and Japan)?

Phase III - Deepening of the perspective of the informal caregivers:

3a) What experiences do informal caregivers have of people with dementia's use of time assistive products in daily situations? 3b) How does this use affect the situation of informal caregivers?

Procedure and data Collection

As the primary outcome measures Kit for Time-processing ability (KaTid), Self-rating of daily time management (Time-S) and Time-Proxy scale for rating daily time management (Time-P) have not been used for the target group, the instruments and the procedure of the assessments have been evaluated by experienced occupational therapists working with persons with dementia. The instruments and the procedure of the assessments have been adapted for different cultural contexts in Sweden, India and Japan".

The recruited PwDs will be randomly allocated to an intervention group or a control group.

All PwD, both randomized to intervention group and to waiting/control group, will have an information brochure about daily time management, frequent problems, and suggested strategies to manage them.

Main assessment points will be at baseline, three months post-baseline and six months post-baseline.

The intervention group will receive a time assistive product as support in daily time management. The time assistive product will be prescribed and introduced by the occupational therapist that identified the participant. The control group will receive a time assistive product after 3 months.

The assessments and interviews with persons with dementia and an informal caregiver will be conducted in the memory clinic, or in the participants' homes, depending on what the persons with dementia and their informal caregivers prefer. Assessments and interviews will be performed first with PwD and then with their informal caregiver.

Data Analysis

Quantitative data will be analyzed using SPSS (Version 23 or later) for Windows, with descriptive, bivariate and multivariable analyses as appropriate performed in order to determine both significant differences between intervention and control group in primary outcomes (daily time management, well-being, COPE Index), significant changes over time within the intervention group, and within/between group interaction effects. Analyses will also be conducted to explore the strength and directions of the relationships between variables in figure 1 in order to arrive at an empirically based model.

Qualitative analysis of data from focus group interviews (I) and individual interviews (Phase III) will be performed using qualitative content analysis inspired by Graneheim and Lundman (2004). The material will be processed by a verbatim transcription, and thoroughly analysed in relation to the research questions posed.

This protocol for registration will focus only on the Phase II, Intervention with focus on persons with dementia and their informal caregivers, the randomized and controlled study, research questions 2a-2d.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate dementia (as determined by MMSE or CDR score)
* Self-rated difficulties in daily time management or difficulties identified by caregivers.
* The person with dementia should know of their disease and feel comfortable discussing experiences related it.
* The persons should be interested in trying out an assistive product as support in everyday activities for a six-month period.
* For each person with dementia, one informal caregiver involved in providing support to the person with dementia (PwD), will be included.

Exclusion Criteria:

* Severe Dementia, ≤ 9 MMSE
* Mental health problems or psychiatric disorders not connected to dementia status,
* High levels of physical frailty,
* Inability to communicate verbally

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Canadian Occupational Performance Measure (COPM) | 3 months
  COPM is used to identify and measure performance and satisfaction with performance of activities that are meaningful and important for the person with dementia to be able to carry out with support of an assistive product. The one - three prioritized activities are rated on a scale ranging from 1 to 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction. COPM was used for persons with Alzheimers disease and can measure change (Clare et al 2010). Change over time in performance and satisfaction with performance on each activity are deemed to be clinically significant when a change of >2 points occurs (Lindqvist et al., 2013).
Change from baseline in Kit for Time-processing ability (KaTid) | 3 months
  KaTid is a standardized and validated instrument. The items, ranging from easy to hard items, in a flip-page format, most items with pictures to make the instrument accessible for people with cognitive and physical disabilities. The instrument operationalizes the concepts of International Classification of Functioning (ICF): Time perception, time orientation and time management. The items in time perception compare the duration of everyday activities. The items measuring time orientation locating today, time concepts, telling time and quantity of time. The items in time management includes questions about what one would have time to do in a set period, when and for how long to do it. The KaTid in original has good psychometric properties (Cronbach's alpha.78 - .86) (Janeslätt, 2012can be used to evaluate interventions (Wennberg et al., 2018). In this study, a short version with 29 items that fit the capacity of people with mild or moderate dementia will be used.

SECONDARY OUTCOMES:
Change from baseline in Time-Selfrating (Time-S) | 3 months
  Self-rating of daily time management; evaluated in adults with psychiatric and neuropsychiatric disabilities and was found to have acceptable psychometric properties (Janeslätt et al., 2015).
Change from baseline in Time-Proxy | 3 months
  Time-Proxy is a proxi-rating for caregivers rating the daily time management of the person with Dementia. A version for parents rating the daily time management of children with similar questions had acceptable psychometric properties (Cronbach Alpha of 0.79 - 0.86) and was used as primary outcome in an randomized controlled study with positive results (Wennberg et al., 2017).
Change from baseline in World Health Organisation Well-being Index (WHO-5) | 3 months
  WHO-5 will be used to measure well-being (Heun et al., 2001), a five item scale producing a score range of 0-25, with higher scores indicating greater psychological well-being.
Change from baseline in Carers of Older People in Europe (COPE) Index | 3 months
  COPE Index (Balducci et al., 2008), measuring negative impact of care, positive value of care, and quality of support
Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (Quest) | 3 months
  Quest 2.0 is used to evaluate user satisfaction of an assistive product. The questionnaire consists of 12 items. A scale ranging from 1 to 5 is used, where 1 indicates not satisfied at all with the device and 5 very satisfied with the device.
Demographic data | Baseline
  A study specific questionnaire of demographic data including age, gender, caregiving characteristics and circumstances, country, cultural features (e.g., mono/polychronic) etc.) will be collected from the PwD and from the informal caregiver.

OTHER OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline
  From patient records to know level of Dementia; mild or moderate.
Clinical Dementia Rating Worksheet (CDR) | Baseline
  From patient records to know level of Dementia; mild or moderate.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnel Janeslätt, PhD, Principal Investigator — Centre for Clinical Research Dalarna, Nissers väg 3, SE-791 82 Falun, Sweden
Locations (1):
- Center fro Clinical Research in Dalarna, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janeslatt G, Lindstedt H, Adolfsson P. Daily time management and influence of environmental factors on use of electronic planning devices in adults with mental disability. Disabil Rehabil Assist Technol. 2015;10(5):371-7. doi: 10.3109/17483107.2014.917124. Epub 2014 May 8. PMID 24805929
- [Background] Boman IL, Nygard L, Rosenberg L. Users' and professionals' contributions in the process of designing an easy-to-use videophone for people with dementia. Disabil Rehabil Assist Technol. 2014 Mar;9(2):164-72. doi: 10.3109/17483107.2013.769124. Epub 2013 Apr 23. PMID 24512219
- [Background] Balducci C, Mnich E, McKee KJ, Lamura G, Beckmann A, Krevers B, Wojszel ZB, Nolan M, Prouskas C, Bien B, Oberg B. Negative impact and positive value in caregiving: validation of the COPE index in a six-country sample of carers. Gerontologist. 2008 Jun;48(3):276-86. doi: 10.1093/geront/48.3.276. PMID 18591353
- [Background] Clare L, Linden DE, Woods RT, Whitaker R, Evans SJ, Parkinson CH, van Paasschen J, Nelis SM, Hoare Z, Yuen KS, Rugg MD. Goal-oriented cognitive rehabilitation for people with early-stage Alzheimer disease: a single-blind randomized controlled trial of clinical efficacy. Am J Geriatr Psychiatry. 2010 Oct;18(10):928-39. doi: 10.1097/JGP.0b013e3181d5792a. PMID 20808145
- [Background] Lindqvist E, Larsson TJ, Borell L. Experienced usability of assistive technology for cognitive support with respect to user goals. NeuroRehabilitation. 2015;36(1):135-49. doi: 10.3233/NRE-141201. PMID 25547777
- [Background] Lindqvist E, Nygard L, Borell L. Significant junctures on the way towards becoming a user of assistive technology in Alzheimer's disease. Scand J Occup Ther. 2013 Sep;20(5):386-96. doi: 10.3109/11038128.2013.766761. Epub 2013 Feb 11. PMID 23394183
- [Background] Wennberg B, Janeslatt G, Kjellberg A, Gustafsson PA. Effectiveness of time-related interventions in children with ADHD aged 9-15 years: a randomized controlled study. Eur Child Adolesc Psychiatry. 2018 Mar;27(3):329-342. doi: 10.1007/s00787-017-1052-5. Epub 2017 Sep 27. PMID 28956183
- [Background] Arntzen C, Holthe T, Jentoft R. Tracing the successful incorporation of assistive technology into everyday life for younger people with dementia and family carers. Dementia (London). 2016 Jul;15(4):646-62. doi: 10.1177/1471301214532263. Epub 2014 Apr 29. PMID 24784941